CLINICAL TRIAL: NCT00956085
Title: Open -Label Trial on the Effects of Memantine in Adults With Obsessive-Compulsive Disorder After a Single Ketamine Infusion
Brief Title: Memantine Augmentation in Treatment-Resistant Adults With Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6924R/5972
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Experimental): Open label memantine titrated in 5mg increments weekly to target dose of 10mg po bid for up to 6 weeks. Memantine was continued to 12 weeks in those with treatment response,13 either previous response to ketamine (≥ 35% Y-BOCS reduction 1 week after IV ketamine) or current response to memantine (≥ 35% Y-BOCS reduction from pre- to post-6 weeks of memantine).
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Open label memantine titrated in 5mg increments weekly to target dose of 10mg po bid for up to 6 weeks. Memantine was continued to 12 weeks in those with treatment response,13 either previous response to ketamine (≥ 35% Y-BOCS reduction 1 week after IV ketamine) or current response to memantine (≥ 35% Y-BOCS reduction from pre- to post-6 weeks of memantine).
  Other Names: Namenda

SUMMARY:
Obsessive-compulsive disorder (OCD) is a common psychiatric illness that affects up to 2-3% of the population. People with OCD experience anxiety-provoking, intrusive thoughts, known as obsessions, and feel compelled to perform repetitive behaviors, or compulsions. The only medications proven effective for OCD are serotonin reuptake inhibitors (SRIs), but even with SRI treatment, most patients continue to experience significant OCD symptoms, impaired functioning, and diminished quality of life. Recent evidence suggest that a different neurotransmitter, glutamate, may contribute to the symptoms in OCD. Medications that target glutamate hold promise for ameliorating symptoms for those patients continuing to suffer from OCD. In this study the investigators are recruiting patients to receive the drug memantine, which is thought to modulate the neurotransmitter glutamate, added to whatever other OCD medications they are taking.

Open label memantine will be titrated in 5mg increments weekly to target dose of 10mg po bid for up to 6 weeks. Memantine will be continued to 12 weeks in those with treatment response,13 either previous response to ketamine (≥ 35% Y-BOCS reduction 1 week after IV ketamine) or current response to memantine (≥ 35% Y-BOCS reduction from pre- to post-6 weeks of memantine).

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Primary Diagnosis of OCD
3. Physically healthy and females must be using effective contraception
4. At lease moderate OCD symptoms (Yale-Brown Obsessive-Compulsive Scale [YBOCS]score greater or equal to 16 prior to entering trial)
5. Able to provide consent
6. May be on or off selective reuptake inhibitor (SRI) medications

   1. Patients on an SRI medication will be included if the dose is stable and adequate (or if they don't want to increase their dose [e.g. side effects] and have a history of prior SRI or CBT treatment meeting criteria for adequate trial)
   2. Patients not on an SRI medication will be included if they they have failed at least 1 prior trial of standard OCD treatment (e.g. SRIs or CBT)

Exclusion Criteria:

1. Ongoing treatment with memantine
2. Patients planning to start CBT during the study period or those who have started CBT within 8 weeks prior to study enrollment
3. Presence of psychotic symptoms or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder.
4. Current major depressive disorder (patients must be free of the disorder for three months prior to enrollment). Patients will be excluded if they are moderately to severely depressed, but if they are mildly to moderately depressed they will be included (Hamilton Depression Rating Scale must be <18).
5. Judged clinically to be at risk of suicide (suicidal ideation, severe depression, or other factors).
6. Current eating disorder
7. Females who are pregnant or nursing
8. Severe renal insufficiency, severe hepatic impairment, or seizure disorder.
9. Documented history of hypersensitivity or intolerance to memantine.
10. Concomitant use of trimethoprim, N-methyl-D-aspartate receptor medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I Rodriguez, M.D., Ph.D., Principal Investigator — Stanford University; Helen B Simpson, MD, PhD, Principal Investigator — NYSPI-Columbia
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodriguez CI, Levinson A, Zwerling J, Vermes D, Simpson HB. Open-Label trial on the effects of memantine in adults with obsessive-compulsive disorder after a single ketamine infusion. J Clin Psychiatry. 2016 May;77(5):688-9. doi: 10.4088/JCP.15l10318. No abstract available. PMID 27249077
- See also: Columbia University Obsessive-Compulsive Disorder Research Clinic — http://www.columbia-ocd.org/
- See also: Rodriguez Lab - Stanford University — http://rodriguezlab.stanford.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Memantine
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Yale-Brown Obsessive-Compulsive Scale.
Description: Patients given YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response was defined as at least a 35% reduction on the YBOCS.
Time Frame: Baseline and 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Memantine: Open label memantine titrated in 5mg increments weekly to target dose of 10mg po bid for up to 6 weeks. Memantine was continued to 12 weeks in those with treatment response, either previous response to ketamine (≥ 35% Y-BOCS reduction 1 week after IV ketamine) or current response to memantine (≥ 35% Y-BOCS reduction from pre- to post-6 weeks of memantine).
Arm/Group | Memantine
Number analyzed (Participants) | 12
Participants | 4

ADVERSE EVENTS:
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=12)
Dizziness (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No